CLINICAL TRIAL: NCT07214259
Title: Development and Testing of an Integrated Care Coordination Intervention for Alcohol Use Disorder Recovery After Liver Transplantation
Brief Title: Intervention for Alcohol Use Disorder Recovery After Liver Transplantation
Acronym: ILTARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh Anne Dageforde (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Leigh Anne Dageforde, Associate Professor of Surgery, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 251447; K23AA031068 (NIH)
Record Dates: First submitted 2025-09-24; First posted 2025-10-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Liver Transplant Recipient; Alcohol Use Disorders (AUD)
Keywords: liver transplant; alcohol use disorder; alcohol associated liver disease; recovery coach; sober active community
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The participants in the control arm will work with a recovery coach and have weekly phone calls with the recovery coach. They will visit the clinic every 3 months for an in-person visit and to complete survey measures related to the study.
  Interventions: Behavioral: Recovery coach
- Intervention (Experimental): The participants in the intervention arm will work with a recovery coach and have weekly phone calls with the recovery coach. They will also have access to an online sober active community that they can use to augment their recovery process. They will visit the clinic every 3 months for an in-person visit and to complete survey measures related to the study.
  Interventions: Behavioral: Online Sober Active Community; Behavioral: Recovery coach

INTERVENTIONS:
Behavioral: Online Sober Active Community — Participants will have access to an online sober active community that they can use to augment their recovery process.
  Arms: Intervention
Behavioral: Recovery coach — Participants will work with a recovery coach including having weekly phone calls with that recovery coach.

SUMMARY:
The goal of this clinical trial is to learn if it is feasible and acceptable to use a recovery coach and an online sober active community to help with alcohol use disorder after liver transplant. The main questions it aims to answer are:

* Is using a recovery coach after liver transplant to help with alcohol use recovery feasible and acceptable?
* Is using an online sober active community after liver transplant to help with alcohol use recovery feasible and acceptable? Researchers will compare standard of care including a recovery coach alone to a recovery coach plus to assist with recovery from alcohol use recovery after liver transplant

Participants will:

* Work with a recovery coach including a weekly phone call
* Visit the clinic once every 3 months for a checkup and to complete surveys
* If randomized to the intervention arm, download an online application with access to a digital sober active community

DETAILED DESCRIPTION:
Rates of alcohol use disorder and alcohol associated liver disease requiring liver transplantation continue to rapidly rise. Return to alcohol use after liver transplant is associated with increased rates of liver transplant failure and mortality, but there is no evidence-based integrated intervention to address alcohol use disorder in liver transplant recipients. The goal of this pilot feasibility randomized control trial is to address a critical gap in knowledge and care for liver transplant recipients with concurrent alcohol use disorder by developing and pilot testing an integrated liver transplant and alcohol recovery program (ILTARP) consisting of a recovery coach supporting post-transplant alcohol relapse prevention, outreach, and care coordination with the added intervention of access to an active sober community. The investigators will conduct a pilot feasibility study of the newly developed ILTARP intervention testing feasibility, acceptability, and potential effectiveness of ILTARP in the liver transplant clinical setting.

ELIGIBILITY:
Inclusion Criteria for Enrollment:

* Age greater than or equal to 21 years old
* Recipient of liver transplant less than or equal to 5 years ago
* History of alcohol use disorder
* Able to understand the purpose of the study and willing to participate and sign informed consent
* Has a smart phone to use for contact with recovery coach and the digital sober active community without additional personal cost
* Willing to participate in online digital community

Exclusion Criteria for Enrollment

* Liver transplant recipient for reason other than alcohol associated liver disease
* Liver transplant greater than 5 years ago
* No mechanism for regular phone contact
* No ability to utilize an application for a digital sober active community
* Any condition that in the opinion of the PI introduces undue risk by participating in this study
* less than 21 years of age
* no history of alcohol use disorder
* Any condition that in the opinion of the PI introduces undue risk by participating in this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of ILTARP (The perception that ILTARP is palatable, agreeable, or satisfactory) | Baseline, month 3, month 6, month 9, and study end (1 year)
  Measured by the Acceptability of Intervention Measure (AIM) survey. The scale ranges from 3 to 15 with a high score indicating greater acceptability.
Feasibility of ILTARP (the degree to which ILTARP can be carried out successfully) | Baseline, month 3, month 6, month 9, and study end (1 year)
  Measured by the Feasibility of Intervention Measure (FIM) survey. The scale ranges from 3 to 15 with a high score indicating greater feasibility.
Appropriateness of ILTARP (ILTARP suitability and relevance) | Baseline, month 3, month 6, month 9, and study end (1 year)
  Measured by the Intervention Appropriateness Measure (IAM).The scale ranges from 3 to 15 with a high score indicating greater appropriateness.

SECONDARY OUTCOMES:
Alcohol use clinically based on lab | Baseline, month 3, month 6, month 9, and study end (1 year)
  the lab test phosphatidylethanol will be used to assess alcohol use
Alcohol use based on self report | Baseline, month 3, month 6, month 9, and study end (1 year)
  Alcohol use will be self reported using the Alcohol Use Disorders Identification (AUDIT-C) scale. The scale ranges from 0 to 12 with 0 being the lowest amount of alcohol and 12 being the most amount of alcohol.
Alcohol cravings based on self report | Baseline, month 3, month 6, month 9, and study end (1 year)
  Alcohol cravings will be self reported using the Penn Alcohol Craving Scale (PACS). Scale score ranges from 0-30 with 0 being the least amount of cravings and 30 the most.
engagement in recovery resources | Baseline, month 3, month 6, month 9, and study end (1 year). The participants will select what resources they have used and how often they have been used. This is not a summarized scale therefore there is not a better or worse outcome.
  Participants will complete a survey on their engagement in recovery resources.
clinic and lab adherence | Baseline, month 3, month 6, month 9, and study end (1 year)
  The number of missed lab appointments and transplant clinic no-show rates will be calculated from the medical record.
medication adherence | Baseline, month 3, month 6, month 9, and study end (1 year)
  Tacrolimus levels will be obtained from the medical record to calculate tacrolimus intrapatient variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All PID that underlie results in a publication can be shared with proper requests.
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: This de-identified data will be available through the NIH mandatory data share through the National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAA-DA). Requests for data sharing will be directed to the NIAAA-DA as the primary mechanism to obtain data.
  If unable to be obtained through the NIAAA-DA, a written proposal maybe submitted with planned analyses and use of the data. Each proposal will be reviewed. Only completely de-identified data will be shared. The recipient of the data must have institutional review board approval. There must be an approved and signed data use agreement.
URL: https://nda.nih.gov/niaaa